CLINICAL TRIAL: NCT03006861
Title: Randomized, Double-blind, Placebo-controlled, Short Term Trial of DelivraTM Livsport Preworkout Cream With or Without Oral Creatine for Improved Power Output and Reduction of Muscle Fatigue During Resistant Training
Brief Title: Delivra Topical Creatine Combined With Oral Creatine for Improving Muscular Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Guelph (Other); University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-145b
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral creatine supplementation (Experimental): 21 g/d oral creatine for 7 days
  Interventions: Dietary Supplement: 3.5 mL/d topical creatine; Dietary Supplement: 3.5 mL/d topical placebo; Dietary Supplement: 21 g/d Oral creatine
- Oral placebo supplementation (Placebo Comparator): 21 g/d oral placebo for 7 days
  Interventions: Dietary Supplement: 3.5 mL/d topical creatine; Dietary Supplement: 3.5 mL/d topical placebo; Dietary Supplement: 21 g/d oral placebo

INTERVENTIONS:
Dietary Supplement: 3.5 mL/d topical creatine
Dietary Supplement: 3.5 mL/d topical placebo
Dietary Supplement: 21 g/d Oral creatine
  Arms: Oral creatine supplementation
Dietary Supplement: 21 g/d oral placebo
  Arms: Oral placebo supplementation

SUMMARY:
Creatine is a nutritional supplement that is often ingested to improve exercise performance. The advent of a new product that is applied to the skin overlying muscle offers potential benefit, if the creatine can be targeted to specific muscles. The investigators are testing a novel creatine cream to determine the effects on human muscular performance. The investigators are assessing whether 7 days of topical creatine application is additive to orally-ingested creatine for improving muscular power (determined by knee extension).

DETAILED DESCRIPTION:
Creatine monohydrate is a popular nutritional supplement with athletes involved in sports involving strength and power. When creatine is orally ingested it combines with inorganic phosphate to form phorylcreatine (PCr) in skeletal muscle . Adenosine Triphosphate (ATP) is the immediate source of energy in muscle - during exercise ATP is broken down to Adenosine Diphosphate (ADP) and inorganic phosphate. Duration of high-intensity exercise is limited to a few seconds based on limited ATP stores in muscle. PCr acts to re-phosphorylate ADP to form ATP so that muscle contraction can continue at high intensities. After creatine monohydrate is ingested, high-intensity exercise capacity is increased because of the increased PCr stores in muscle.

Traditionally, creatine is consumed orally as a supplement. Delivra Inc. has developed a topical cream containing creatine that is designed to penetrate the skin. The study purpose is to determine whether topically-applied creatine is additive with orally-ingested creatine for improving muscular strength and power.

The hypothesis is that topically-applied creatine is additive with orally-ingested creatine for improving muscular performance.

The study involves a double-blind placebo-controlled parallel group design. Participants (n=132) will be randomized to receive either oral creatine supplementation or placebo (21 g/d) for 7 days. One leg of each participant will be randomized to receive topical creatine (3.5 mL/d) and the opposite leg placebo for 7 days.

The baseline assessment involves measuring muscular power during 5 sets of 15 repetitions of knee extension on a dynamometer, with each set separated by 1 minute rest, with each leg tested separately. Additional measures include assessment of body composition and body water content. Participants will then receive either oral creatine (21 g/d) or placebo for 7 days. One leg of each participant will be randomized to receive topical creatine (3.5 mL/d) and the opposite leg placebo for 7 days. The same assessments as done at baseline will then be repeated after the 7 days of creatine supplementation.

The primary outcomes are average and peak power output.

ELIGIBILITY:
Inclusion Criteria:

* Physically active and able to pass Physical Activity Readiness Questionnaire

Exclusion Criteria:

* Allergies to any ingredients in the cream
* Answering "yes" to Physical Activity Readiness Questionnaire
* Currently pregnant or breastfeeding,
* Presence of significant medical disorder that would compromise the participant's safety to take part in the trial (eg: cancer, immunosuppressed)
* History of alcohol or drug abuse within the past year
* Anyone using recreational drugs
* Use of performance enhancing drugs or supplements within 2 months including caffeine and creatine in supplement form
* Currently using other topical agents for treatment of pain or inflammation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in average power across 5 set of 15 repetitions separated by 60s rest on an isokinetic dynamometer | Change from baseline to 7 days

SECONDARY OUTCOMES:
Change in body composition (percent fat) | Change from baseline to 7 days
Change in body water content | Change from baseline to 7 days
Change in peak power across 5 set of 15 repetitions separated by 60s rest on an isokinetic dynamometer | Change from baseline to 7 days
Adverse events recorded on adverse event forms | Change from baseline to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, PhD, Principal Investigator — University of Saskatchewan; Jamie Burr, PhD, Principal Investigator — University of Guelph; Travis Saunders, PhD, Principal Investigator — University of Prince Edward Island
Locations (3):
- Canada (3):
  - University of Guelph, Guelph, Ontario
  - University of Prince Edward Island, Charlottetown, Prince Edward Island
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No